CLINICAL TRIAL: NCT03139916
Title: Phase II Clinical Trial of Bavituximab With Radiation and Temozolomide for Patients With Newly Diagnosed Glioblastoma
Brief Title: Bavituximab With Radiation and Temozolomide for Patients With Newly Diagnosed Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Peregrine Pharmaceuticals (Industry); National Comprehensive Cancer Network (Network)
Responsible Party: Principal Investigator, Elizabeth R. Gerstner, MD, Principle Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-037
Record Dates: First submitted 2017-05-02; First posted 2017-05-04 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Glioblastoma
Keywords: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide; bavituximab; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bavituximab + Standard of Care Radiation + Temozolomide (Experimental): Cycle 1 consists of 6 weeks (42 days) of chemoradiation. Radiation therapy is administered per standard of care. Bavituxumab 3 mg/kg IV administration starts during the 1st week of chemoradiation and continues weekly. Temozolomide 75/m2 is administered orally once daily.
  Cycle 2 is 4 weeks (28 days) long and Bavituxumab 3 mg/kg IV administration occurs weekly.
  Cycle 3 and beyond are each 4 weeks (28 days) long. Bavituxumab 3 mg/kg IV administration occurs weekly for a cumulative total of 18 weeks; treatment may continue beyond 18 weeks at the discretion of the treating physician if the participant is deriving clinical benefit. Temozolomide 150-200 mg/m2 is administered orally once daily on days 1-5 in cycles 3 and 4.
  Interventions: Drug: Temozolomide; Drug: Bavituximab; Radiation: Radiation

INTERVENTIONS:
Drug: Temozolomide — Temozolomide causes cell death and shrinks and kills the cancer cells
  Other Names: Temodar
Drug: Bavituximab — Bavituximab may activate (cause) the immune system to attack the cancer cells
Radiation: Radiation — Radiation causes cell death and shrinks and kills the cancer cells.

SUMMARY:
This research study is studying a combination of drugs with radiation as a possible treatment for Glioblastoma.

The drugs involved in this study are:

* Bavituximab
* Temozolomide

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved Bavituximab as a treatment for any disease.

The FDA has approved Temozolomide as a treatment option for this disease.

In this research study, the investigators are studying how the combination of Bavituximab, Temozolomide, and radiation affects this cancer. The current standard care of treatment for newly diagnosed glioblastoma is the combination of Temozolomide and radiation. Temozolomide causes cell death and radiation shrinks and kills the cancer cells. Bavituximab may activate (cause) the immune system to attack the cancer cells as well as target tumor cells themselves to kill them.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed newly diagnosed glioblastoma or glioblastoma variant (ex. gliosarcoma), including documentation of unmutated isocitrate dehydrogenase (IDH) by immunohistochemistry (sequencing not required).
* Participants must have 1-4 cm2 measurable disease (4 cm2 is the maximal size). See Section 11 for the evaluation of measurable disease. Disseminated GBM is not allowed.
* No prior immunotherapy allowed or prior alkylating agents or prior radiation to the brain.
* Age >17 years since adult GBM is biologically different from pediatric GBM and there is no data for bavituximab in pediatric populations.
* Karnofsky ≥60%, see Appendix A
* Life expectancy of greater than 6 months.
* Participants must have normal organ and marrow function as defined below:

  * leukocytes ≥3,000/mcL
  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * total bilirubin within normal institutional limits (unless patient has Gilbert's syndrome in which total bilirubin should be ≤ 2xULN)
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
  * creatinine within normal institutional limits OR
  * creatinine clearance ≥60 mL/min/1.73 m2 for participants with creatinine levels above institutional normal(using Cockcroft Gault Formula)
  * negative serum pregnancy test in WOCBP
  * INR/PT ≤1.5 x institutional ULN unless subject is receiving anticoagulant therapy as long as PT or INR is within therapeutic range of intended use of anticoagulants
  * aPTT ≤1.5 x institutional ULN unless subject is receiving anticoagulant therapy as long as PTT is within therapeutic range of intended use of anticoagulants
* < 4 mg dexamethasone daily (or equivalent if on another corticosteroid) at time of start of therapy. Patients on a steroid taper post-surgery and are anticipated to be on <4 mg at time of chemoradiation initiation will be eligible to consent but to initiate treatment on trial, the participant must be on <4 mg or equivalent of steroids otherwise participate will be deemed a screen fail and be replaced.
* The effects of bavituximab on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of bavituximab administration.
* Able to undergo an MRI scan and receive gadolinium-based contrast.
* 1 cm3 of available tissue.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Participants who are receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to bavituximab.
* Participants receiving any medications or substances that are moderate and/or potent enzyme inducers or inhibitors which may have an effect on the metabolism of bavituximab. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product (Appendix C for partial list).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because bavituximab is an immunotherapy agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with bavituximab breastfeeding should be discontinued if the mother is treated with bavituximab. These potential risks may also apply to other agents used in this study.
* HIV-positive participants on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with bavituximab. In addition, these participants are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.
* Participants with other active malignancy in the past 3 years excluding in situ tumors.
* Participants must meet the following windows from procedures (there is no window required for port placement since there is no anticipated impact on wound healing with bavituximab):

  * Major surgery (ex. craniotomy) within 3 weeks of initiation of treatment.
  * Brain biopsy within 2 weeks
* Participants with history of bleeding disorder/coagulopathy.
* Participants with history of chronic or acute hepatitis C or B infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth R Gerstner, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts general Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ly KI, Richardson LG, Liu M, Muzikansky A, Cardona J, Lou K, Beers AL, Chang K, Brown JM, Ma X, Reardon DA, Arrillaga-Romany IC, Forst DA, Jordan JT, Lee EQ, Dietrich J, Nayak L, Wen PY, Chukwueke U, Giobbie-Hurder A, Choi BD, Batchelor TT, Kalpathy-Cramer J, Curry WT, Gerstner ER. Bavituximab Decreases Immunosuppressive Myeloid-Derived Suppressor Cells in Newly Diagnosed Glioblastoma Patients. Clin Cancer Res. 2023 Aug 15;29(16):3017-3025. doi: 10.1158/1078-0432.CCR-23-0203. PMID 37327319

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bavituximab + Standard of Care Radiation + Temozolomide
Started | 36
Completed | 33
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Clinical progression prior to start of study treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bavituximab + Standard of Care Radiation + Temozolomide
Number analyzed (Participants) | 33
Age, Continuous [Mean (Full Range); unit: years] | 59 [24 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 32
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival at 12 Months (OS12)
Description: Overall survival is defined as the time from study entry to death from any cause. OS12 is the percentage of subjects who are alive 12 months after study entry. Data for subjects who are lost to follow up prior to documented death will be counted as deaths at the last assessment date when the subject is known to be alive.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bavituximab + Standard of Care Radiation + Temozolomide
Number analyzed (Participants) | 33
percentage of participants | 72.7 [59 to 90]

2. Secondary Outcome: Radiographic Response Rate
Description: Radiographic response (RR) is defined as a complete response or partial response per RANO (Response assessment in neuro-oncology) criteria with incorporation of iRANO (immunotherapy response assessment for neuro-oncology) criteria. The radiographic response rate is the percentage of subjects who achieved radiographic response as defined above.
Time Frame: every 3 months for 5 years
Population: Out of 33 patients, 26 patients had measurable disease at baseline per RANO criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Bavituximab + Standard of Care Radiation + Temozolomide
Number analyzed (Participants) | 26
Participants | 4

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival is defined as the time of study entry to time of disease progression, or death due to any cause. Data for subjects who are lost to follow up will be censored at the date when the subject is last known to be alive. PFS results below are reported up to the data cutoff in May 2021.
Time Frame: every 3 months for up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Bavituximab + Standard of Care Radiation + Temozolomide: * Bavituximab will be administered weekly intravenously
  * Temozolomide will be administered daily
  * Standard of Care Radiation will be administered per hospital guideline.
  Temozolomide: Temozolomide causes cell death and shrinks and kills the cancer cells
  Bavituximab: Bavituximab may activate (cause) the immune system to attack the cancer cells
  Radiation: Radiation causes cell death and shrinks and kills the cancer cells.
Arm/Group | Bavituximab + Standard of Care Radiation + Temozolomide
Number analyzed (Participants) | 33
months | 6.9 [6.2 to 9.7]

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time of study entry to death from any cause. Data for subjects who are lost to follow up will be censored at the date when the subject is last known to be alive. OS results below are reported up to the data cutoff in May 2021.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bavituximab + Standard of Care Radiation + Temozolomide
Number analyzed (Participants) | 33
months | 15.4 [13.3 to 23.6]

ADVERSE EVENTS:
Time Frame: Up to 5 years, starting at date of first treatment administration.
Arm/Group | Bavituximab + Standard of Care Radiation + Temozolomide
All-Cause Mortality (participants affected / at risk) | 29/36
Serious Adverse Events (participants affected / at risk) | 9/36
Other Adverse Events (participants affected / at risk) | 33/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bavituximab + Standard of Care Radiation + Temozolomide (N=36)
Cognitive disturbance (Nervous system disorders) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Methicillin-Sensitive Staphylococcus aureus Ventricular Shunt Infection
Hydrocephalus (Nervous system disorders) | 2
Nervous system disorders - Other, specify (Nervous system disorders) | 1 — Altered Mental Status
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 — Obstructive pyelonephritis
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 — Aspiration Pneumonia
Somnolence (Nervous system disorders) | 2
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 — Bilateral lower extremity DVTs
Confusion (Psychiatric disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 1 — L. Binocular Horizontal Diplopia
Fever (General disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 1 — DVT
Headache (Nervous system disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 3
Skin/subcutaneous tissue disorders; Other, specify (Skin and subcutaneous tissue disorders) | 1 — Varicella Zoster Infection
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bavituximab + Standard of Care Radiation + Temozolomide (N=36)
Abdominal pain (Gastrointestinal disorders) | 3
Agitation (Psychiatric disorders) | 2
Akathisia (Nervous system disorders) | 1
Alanine aminotransferase increased (Investigations) | 9
Alkaline phosphatase increased (Investigations) | 1
Allergic reaction (Immune system disorders) | 1 — Allergy to Naloxene
Alopecia (Skin and subcutaneous tissue disorders) | 12
Anemia (Blood and lymphatic system disorders) | 6
Anorexia (Metabolism and nutrition disorders) | 9
Anxiety (Psychiatric disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Aspartate aminotransferase increased (Investigations) | 9
Ataxia (Nervous system disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3
Bladder spasm (Renal and urinary disorders) | 1
Blood bilirubin increased (Investigations) | 2
Blurred vision (Eye disorders) | 4
Cardiac disorders - Other, specify (Cardiac disorders) | 3 — Tachycardia
Cardiac disorders - Other, specify (Cardiac disorders) | 1 — Elevated Blood Pressure
Cognitive disturbance (Nervous system disorders) | 4
Colonic ulcer (Gastrointestinal disorders) | 2
Concentration impairment (Nervous system disorders) | 2
Confusion (Psychiatric disorders) | 5
Conjunctivitis infective (Infections and infestations) | 1
Constipation (Gastrointestinal disorders) | 23
Cough (Respiratory, thoracic and mediastinal disorders) | 5
CPK increased (Investigations) | 1
Creatinine increased (Investigations) | 1
Cushingoid (Endocrine disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 6
Delirium (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 3
Diarrhea (Gastrointestinal disorders) | 6
Dizziness (Nervous system disorders) | 12
Dry eye (Eye disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Duodenal hemorrhage (Gastrointestinal disorders) | 3
Dysgeusia (Nervous system disorders) | 3
Dysmenorrhea (Reproductive system and breast disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 5
Dysphasia (Nervous system disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 — Muffled hearing
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 — Ear Wax Buildup
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 — Left Ear Dryness
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 — Right Ear Skin Irritation
Ear pain (Ear and labyrinth disorders) | 1
Edema cerebral (Nervous system disorders) | 1
Edema limbs (General disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2
External ear pain (Ear and labyrinth disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 1 — Right Ptosis
Eye disorders - Other, specify (Eye disorders) | 1 — Disconjugate Gaze
Eye disorders - Other, specify (Eye disorders) | 1 — Acute Infarct in Right Lentiform Nucleus
Eye disorders - Other, specify (Eye disorders) | 1 — L. upper eyelid stye
Eye disorders - Other, specify (Eye disorders) | 1 — Retinal Hemorrhage
Eye disorders - Other, specify (Eye disorders) | 1 — R. Homonymous Hemianopia
Eye disorders - Other, specify (Eye disorders) | 1 — Vision Issues
Eye disorders - Other, specify (Eye disorders) | 1 — Swollen Eyes
Eye infection (Infections and infestations) | 1
Facial muscle weakness (Nervous system disorders) | 1
Fall (Injury, poisoning and procedural complications) | 3
Fatigue (General disorders) | 27
Fecal incontinence (Gastrointestinal disorders) | 1
Fever (General disorders) | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Floaters (Eye disorders) | 3
Flu like symptoms (General disorders) | 2
Gait disturbance (General disorders) | 7
Gastroesophageal reflux disease (Gastrointestinal disorders) | 5
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 — Loose Stools
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Left Sided Neglect
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Choking
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Impaired balance
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Bilateral Tinea Pedis
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Tooth Fracture and Lip Laceration Secondary to Fall
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Left Proximal Arm Discomfort
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Bilateral Shoulder Pain
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Right-sided facial cellulitis
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Hip discomfort
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Bowel incontinence
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Rash in groin
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Skin Tears on Coccyx
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Erythematous Lesion
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Episode of inability to walk
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Diabetes Mellitus Type 2
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Sleepwalking
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Mouth Sore
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Bad breath/hallitosis
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Oral thrush
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Herpes zoster
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Right Upper Extremity Pronator Drift
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Dysfluent speech
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Word finding difficulty
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Night sweats
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Bilateral leg cramps at night
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Numbness in R. Pinky Finger, Toes, and Left Shin
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Increased thirst
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Bilateral Ankle Swelling
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Right-sided incision pain
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Itching
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Panic Attacks
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5
Growth suppression (Musculoskeletal and connective tissue disorders) | 1 — Right Hand cramping
Headache (Nervous system disorders) | 18
Hematuria (Renal and urinary disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3
Hydrocephalus (Nervous system disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 7
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 4
Infections and infestations - Other, specify (Infections and infestations) | 1 — Propionibacterium acnes infection
Infections and infestations - Other, specify (Infections and infestations) | 1 — Hepatitis
Infections and infestations - Other, specify (Infections and infestations) | 1 — Viral Infection
Infections and infestations - Other, specify (Infections and infestations) | 1 — Cold
Infections and infestations - Other, specify (Infections and infestations) | 1 — Rash
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 — Abrasion
Insomnia (Psychiatric disorders) | 12
Intracranial hemorrhage (Nervous system disorders) | 1
Investigations - Other, specify (Investigations) | 1 — Swollen gums
Investigations - Other, specify (Investigations) | 1 — Suture Wound
Investigations - Other, specify (Investigations) | 1 — Rash
Investigations - Other, specify (Investigations) | 1 — Neutropenia
Investigations (Investigations) | 1 — Cold-like symptpms
Investigations - Other, specify (Investigations) | 1 — Numbness
Investigations - Other, specify (Investigations) | 1 — Elevated d-dimer
Investigations - Other, specify (Investigations) | 1 — Tachycardia
Investigations - Other, specify (Investigations) | 1 — Skin abscess
Investigations - Other, specify (Investigations) | 1 — L. Paravertebral Discomfort
Investigations - Other, specify (Investigations) | 1 — Benign Prostatic Hyperplasia
Investigations - Other, specify (Investigations) | 1 — Word Finding Difficulty
Investigations - Other, specify (Investigations) | 1 — R. Lower Facial Drooping
Investigations - Other, specify (Investigations) | 1 — Lymphopenia
Investigations - Other, specify (Investigations) | 1 — Rigors
Investigations - Other, specify (Investigations) | 1 — Intermittent Left Upward Drift
Investigations - Other, specify (Investigations) | 1 — Intermittent L. Foot Pain
Investigations - Other, specify (Investigations) | 1 — Intermittent Pruritus on Arms and Groin
Investigations - Other, specify (Investigations) | 1 — Eosinophilia
Investigations - Other, specify (Investigations) | 1 — Stomach Cramping
Investigations - Other, specify (Investigations) | 1 — Upward Left Pronator Drift
Investigations - Other, specify (Investigations) | 1 — Worsened Elevated Blood Bilirubin
Irritability (General disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Lip infection (cold sore) (Infections and infestations) | 1
Localized edema (General disorders) | 1
Lymphocyte count decreased (Investigations) | 10
Memory impairment (Nervous system disorders) | 12
Mucosal infection (Infections and infestations) | 1
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 5
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 — Joint Pain
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 — Generalized Pain
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 — Right hand cramping
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Nausea (Gastrointestinal disorders) | 18
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Nervous system disorders - Other, specify (Nervous system disorders) | 1 — Lightheadedness
Nervous system disorders - Other, specify (Nervous system disorders) | 1 — Difficulty Initiating Motor Movements
Nervous system disorders - Other, specify (Nervous system disorders) | 1 — Right facial weakness
Nervous system disorders - Other, specify (Nervous system disorders) | 1 — Migraine
Nervous system disorders - Other, specify (Nervous system disorders) | 1 — Jaw weakness
Nervous system disorders - Other, specify (Nervous system disorders) | 1 — Unable to ambulate-unsteady gait
Nervous system disorders - Other, specify (Nervous system disorders) | 1 — Word Finding Difficulty
Nervous system disorders - Other, specify (Nervous system disorders) | 2 — Word Finding Difficulty
Nervous system disorders - Other, specify (Nervous system disorders) | 1 — Olfactory seizure activity
Nervous system disorders - Other, specify (Nervous system disorders) | 1 — Radicular Nerve Pain
Nervous system disorders - Other, specify (Nervous system disorders) | 1 — Expressive aphasia
Nervous system disorders - Other, specify (Nervous system disorders) | 1 — Intraparenchymal Hemorrhage
Hemiparesis (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Neutrophil count decreased (Investigations) | 8
Non-cardiac chest pain (General disorders) | 1
Nystagmus (Nervous system disorders) | 2
Obesity (Metabolism and nutrition disorders) | 1
Pain (General disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Palpitations (Cardiac disorders) | 1
Papulopustular rash (Infections and infestations) | 2
Paresthesia (Nervous system disorders) | 2
Paronychia (Infections and infestations) | 1
Platelet count decreased (Investigations) | 12
Pruritus (Skin and subcutaneous tissue disorders) | 5
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 — Hypomania
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 — PTSD
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 — Mood alteration
Rash acneiform (Skin and subcutaneous tissue disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 — Difficulty urinating
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 — Nocturia
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 — Chronic Renal Insufficiency
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 — Urine Odor
Seizure (Nervous system disorders) | 8
Sinus bradycardia (Cardiac disorders) | 5
Sinus pain (Nervous system disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Skin/subcutaneous tissue disorders; Other, specify (Skin and subcutaneous tissue disorders) | 1 — Asteatotic Eczema on Left Lower Leg
Skin/subcutaneous tissue disorders; Other, specify (Skin and subcutaneous tissue disorders) | 1 — Livedo Reticularis
Skin/subcutaneous tissue disorders; Other, specify (Skin and subcutaneous tissue disorders) | 1 — Right Eyelid Erythema
Skin/subcutaneous tissue disorders; Other, specify (Skin and subcutaneous tissue disorders) | 1 — basal cell carcinoma on nose
Skin/subcutaneous tissue disorders; Other, specify (Skin and subcutaneous tissue disorders) | 1 — Pruritic Rash
Skin/subcutaneous tissue disorders; Other, specify (Skin and subcutaneous tissue disorders) | 1 — Fungal Infection (ringworm)
Somnolence (Nervous system disorders) | 4
Stomach pain (Gastrointestinal disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 2
Tremor (Nervous system disorders) | 1
Upper respiratory infection (Infections and infestations) | 1
Urinary frequency (Renal and urinary disorders) | 3
Urinary incontinence (Renal and urinary disorders) | 3
Urinary tract infection (Infections and infestations) | 4
Urinary tract pain (Renal and urinary disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Vasovagal reaction (Nervous system disorders) | 1
Vomiting (Gastrointestinal disorders) | 6
Watering eyes (Eye disorders) | 1
Weight gain (Investigations) | 3
Weight loss (Investigations) | 5
White blood cell decreased (Investigations) | 11
Right hemianopsia (Eye disorders) | 1
Myoglobin increase (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/16/NCT03139916/Prot_SAP_000.pdf
  • Informed Consent Form (2019-03-12): https://cdn.clinicaltrials.gov/large-docs/16/NCT03139916/ICF_001.pdf